CLINICAL TRIAL: NCT07360691
Title: Prospective Clinical Evaluation of High-Purity Type I Collagen as a Biologic Reinforcement in Selected High-Risk Hernia Repair Scenarios
Brief Title: Early Clinical Outcomes of High-Purity Type I Collagen as a Biologic Reinforcement in Selected Hernia Repair Scenarios
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/007/2026
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hernia; Ventral Hernia; Incisional Hernia; İnguinal Hernia; Abdominal Wall Hernia; Surgical Site Infection; Postoperative Complications
Keywords: Hernia Repair; Ventral Hernia Repair; Incisional Hernia Repair; Inguinal Hernia Repair; Biological Mesh; Type I Collagen; Wound Healing; Postoperative Pain; Hernia Recurrence
MeSH Terms: conditions — Hernia; Hernia, Ventral; Incisional Hernia; Hernia, Inguinal; Hernia, Abdominal; Surgical Wound Infection; Postoperative Complications; Osteogenesis Imperfecta, Type IV; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPTC-Reinforced Hernia Repair (Experimental): Participants undergo standard hernia repair with primary fascial closure where feasible, reinforced using High-Purity Type I Collagen mesh (Surgicoll-Mesh®). The biologic mesh is used as an adjunct reinforcement and not as a routine replacement for permanent synthetic mesh. Mesh placement (onlay or sublay) and peri-operative management are performed according to surgeon discretion and institutional protocols. The arm evaluates early postoperative safety, wound healing, and short-term clinical outcomes over an 8-week follow-up period in selected high-risk or contaminated hernia repair scenarios.
  Interventions: Device: High-Purity Type I Collagen Mesh

INTERVENTIONS:
Device: High-Purity Type I Collagen Mesh — High-Purity Type I Collagen mesh (>97% purity), un-crosslinked and resorbable, designed to function as a temporary biologic scaffold facilitating host tissue integration and remodeling. The device is applied as a biologic reinforcement following anatomical hernia repair in selected high-risk or contaminated surgical fields where permanent synthetic mesh placement is associated with increased risk.

SUMMARY:
This prospective, single-arm clinical study evaluates the safety, feasibility, and early clinical outcomes of High-Purity Type I Collagen (HPTC; Surgicoll-Mesh®) when used as a biologic reinforcement in selected hernia repair scenarios where permanent synthetic mesh placement is undesirable. Outcomes focus on early postoperative safety, wound healing, and complication profiles over an 8-week follow-up period.

DETAILED DESCRIPTION:
Synthetic mesh has reduced hernia recurrence but is associated with significant complications in contaminated fields and high-risk patients. Biologic meshes offer potential advantages including biocompatibility, resistance to infection, and tissue remodeling. High-Purity Type I Collagen (>97% purity) is an un-crosslinked, resorbable scaffold designed to support host tissue integration.

This prospective observational study systematically evaluates early clinical outcomes following HPTC-reinforced hernia repair, including surgical site infection, wound healing, postoperative pain, and early integrity of repair. The study is not designed to assess long-term recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ventral, incisional, umbilical, or para-umbilical hernia
* Contaminated or potentially contaminated surgical field
* Hernia repair following infected mesh explantation
* High-risk patients (diabetes, obesity, smoking, immunosuppression)
* Ability to provide informed consent

Exclusion Criteria:

* Clean, low-risk primary hernia suitable for synthetic mesh
* Large defects requiring permanent load-bearing prosthesis
* Generalized peritonitis or uncontrolled sepsis
* Known collagen hypersensitivity
* Pregnancy
* Inability to comply with follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Safety and Feasibility | Up to 8 weeks post-operatively
  Incidence of surgical site infection, mesh-related adverse events, and need for re-intervention or mesh removal within 8 weeks following surgery.

SECONDARY OUTCOMES:
Early Wound Healing Outcomes | Up to 8 weeks
  Time to epithelialization, wound complications (seroma, hematoma, dehiscence)
Postoperative Change in Visual Analog Scale (VAS) pain scores | Baseline (preoperatively) to 8 weeks postoperatively
  Change in pain intensity assessed using the Visual Analog Scale for Pain, a patient-reported numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores represent worse pain intensity.
Early Clinical Integrity of Repair | Up to 8 weeks
  Absence of early fascial failure or wound breakdown on clinical examination
Length of Hospital Stay | From immediately after the surgery until hospital discharge
  Number of postoperative inpatient days
Patient Satisfaction With Hernia Repair | 8 weeks post-operatively
  Patient-reported satisfaction with surgical outcome assessed on a 5-point Likert scale:
  Very satisfied / Satisfied / Neutral / Dissatisfied / Very dissatisfied
Hernia-Specific Quality of Life | Baseline and 8 weeks post-operatively
  Hernia-specific quality of life assessed using European Registry for Abdominal Wall Hernias Quality of Life Score (EuraHS-QoL), covering: Pain at rest and during activity, Restriction of activities, Cosmetic discomfort. Scores range from 0 (no impairment) to 90 (worst impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this clinical study will be made available upon reasonable request. Shared data will include baseline characteristics, peri-operative variables, postoperative outcomes, and patient-reported outcome measures collected during the 8-week follow-up period. All shared data will be fully anonymized, with no direct or indirect identifiers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication of the primary study results and will remain available for up to 5 years thereafter.
Access Criteria: Access to de-identified IPD will be granted to qualified researchers upon submission of:
  A methodologically sound research proposal
  Intended use aligned with scientific and ethical standards
  Requests will be reviewed by the study investigators. Data will be shared under a data use agreement to ensure appropriate use and protection of participant confidentiality.

REFERENCES:
- [Background] Arturi K, Harris EJ, Gasser L, Escher BI, Braun G, Bosshard R, Hollender J. MLinvitroTox reloaded for high-throughput hazard-based prioritization of high-resolution mass spectrometry data. J Cheminform. 2025 Jan 31;17(1):14. doi: 10.1186/s13321-025-00950-4. PMID 39891244
- [Background] Ong JEX. How to restore lower complete edentulism with implant-supported overdentures: an evidence-based clinical management. Br Dent J. 2024 Nov;237(10):773-777. doi: 10.1038/s41415-024-7842-5. Epub 2024 Nov 22. PMID 39572811
- [Background] Cevasco M, Itani KM. Ventral hernia repair with synthetic, composite, and biologic mesh: characteristics, indications, and infection profile. Surg Infect (Larchmt). 2012 Aug;13(4):209-15. doi: 10.1089/sur.2012.123. Epub 2012 Aug 22. PMID 22913337
- [Background] Huntington CR, Cox TC, Blair LJ, Schell S, Randolph D, Prasad T, Lincourt A, Heniford BT, Augenstein VA. Biologic mesh in ventral hernia repair: Outcomes, recurrence, and charge analysis. Surgery. 2016 Dec;160(6):1517-1527. doi: 10.1016/j.surg.2016.07.008. Epub 2016 Aug 12. PMID 27528210
- [Background] Cheng AW, Abbas MA, Tejirian T. Outcome of abdominal wall hernia repair with biologic mesh: Permacol versus Strattice. Am Surg. 2014 Oct;80(10):999-1002. PMID 25264647
- [Background] Nahabedian MY, Sosin M, Bhanot P. A Current Review of Biologic Meshes in Abdominal Wall Reconstruction. Plast Reconstr Surg. 2018 Sep;142(3 Suppl):74S-81S. doi: 10.1097/PRS.0000000000004866. PMID 30138272
- [Background] Rhon-Calderon EA, Galarza RA, Lomniczi A, Faletti AG. The systemic and gonadal toxicity of 3-methylcholanthrene is prevented by daily administration of alpha-naphthoflavone. Toxicology. 2016 Apr 15;353-354:58-69. doi: 10.1016/j.tox.2016.05.005. Epub 2016 May 6. PMID 27163632